CLINICAL TRIAL: NCT00414570
Title: An Imaging Study of [18]F-fluoro-3'-Deoxy-3'-L-fluorothymidine ([18]F-FLT) in Patients With Locally Advanced or Metastatic Pancreatic Cancer Who Will be Treated With Gemcitabine or Other Nucleoside Analogs
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Retirement of former Qualified Investigator and lack of resources to complete study
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-FLT-001
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Cancer
Keywords: Positron Emission Tomography (PET); 3'-deoxy-3'(18F)fluorothymidine ([18]F-FLT)
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18]F-FLT PET scan (Experimental): Radioactive dose of 2.59 MBq/kg (range 100 - 350 MBq) [18]F-FLT per injection prior to Positron Emission Tomography (PET) imaging. [18]F-FLT PET scans at baseline/pre-treatment and at disease progression, up to a maximum of two separate [18]F-FLT PET scans per participant.
  Interventions: Drug: [18]F-FLT PET scan

INTERVENTIONS:
Drug: [18]F-FLT PET scan — Injection of [18]F-FLT radiopharmaceutical followed by PET imaging.
  Other Names: [18]F-FLT Positron Emission Tomography scan

SUMMARY:
The objectives of this pilot study are: (i) to compare response to chemotherapy, time to disease progression and overall survival in patients with pancreatic cancer who will be treated with gemcitabine (or other nucleoside analogs) who demonstrate [18]F-FLT uptake to those patients who do not demonstrate [18]F-FLT uptake; (ii) to correlate [18]F-FLT uptake with hENT1 expression in biopsy samples where available; (iii)to determine the presence or absence of uptake, the relative uptake score (RUS), standardized uptake value (SUV), and tumor to background ratios (T/B) of [18]F-FLT in patients with known carcinoma of the pancreas and assess this uptake in relation to time to disease progression; and (iv) to demonstrate the safety of [18]F-FLT.

DETAILED DESCRIPTION:
The proposed clinical trial will be an imaging, open label, non-randomized, single site pilot study in patients with locally advanced or metastatic pancreatic carcinoma who will be treated with gemcitabine or other nucleoside analogs. Study participants will receive an IV injection of 2.59 MBq/kg ± 10% of [18]F-FLT (range: 100 to 350 MBq). If clinically indicated, dynamic PET scan imaging may start immediately before the injection, followed by half-body or limited frame scanning, using either a PET/CT or PET scanner. The first [18]F-FLT PET scan for each subject will occur within 4 weeks prior to commencement of his/her treatment. Study subjects will have a follow-up [18]F-FLT-PET scan at the time of disease progression, to a maximum of two [18]F-FLT PET scans. The same imaging procedure will be followed for both [18]F-FLT PET scans. At the same time as the [18]F-FLT PET scans occur, the patients' index tumour lesions will be re-evaluated by the same imaging modality originally used to assess the index lesions. Images will be interpreted by an experienced Nuclear Medicine physician with regard to normal physiological uptake of [18]F-FLT (RUS, SUV, and T/B). The location and relative uptake of normal and abnormal [18]F-FLT biodistribution patterns will be noted and correlated with time to disease progression and hENT1 expression in biopsy samples, where available. A medical chart review will be done at regular intervals to assess response to treatment, time to disease progression, and overall survival. Disease progression will be determined using the National Cancer Institute's Response Evaluation Criteria In Solid Tumours (RECIST).

ELIGIBILITY:
Inclusion Criteria:

* male or female ≥ 18 years of age. If female of child bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test
* patients with known locally advanced or metastatic carcinoma of the pancreas
* planned gemcitabine treatment
* calculated creatinine clearance >50ml/min (calculated by Crockcraft and Gault equation)
* able and willing to follow instructions and comply with the protocol
* provide written consent prior to participation in this study
* Karnofsky Performance Scale Score 60-100

Exclusion Criteria:

* Bilirubin ≥200 umol/L
* AST or ALT ≥5 times the upper limits of normal
* Serious medical conditions which may prevent a patient from tolerating experimental chemotherapy such as: congestive heart failure, unstable angina, unstable ventricular arrhythmia, uncontrolled psychiatric conditions, serious infections, uncontrolled diabetes
* uncontrolled brain metastasis. Patients who have stable brain metastasis treated with radiation or surgery who are symptomatic and a stable dose of dexamethasone are eligible
* nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
compare response to chemotherapy, time to disease progression and overall survival in pancreatic cancer patients treated with gemcitabine who demonstrate 18F-FLT uptake to those patients who do not demonstrate 18F-FLT uptake | 5 Years
correlate 18F-FLT uptake with hENT1 expression with biopsy samples where available | 5 Years

SECONDARY OUTCOMES:
determine the presence or absence of uptake, the relative uptake score (RUS) and tumor background ratios of 18F-FLT in patients with known carcinoma of the pancreas and assess this uptake in relation to time of disease progression | 5 Years
to demonstrate the safety of 18F-FLT manufactured at the Edmonton PET Centre | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sawyer, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada